CLINICAL TRIAL: NCT03374384
Title: Pattern of Pediatric Seizures at Al-Arish Central Hospital - North Sinai
Brief Title: The Pattern of Pediatric Seizures at Al-Arish Central Hospital - North Sinai
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ehsan M saied (Other)
Responsible Party: Sponsor-Investigator, Ehsan M saied, Assiut, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 17100278
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Convulsive Seizures
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No drug intervention — This study will be performed in Al-Arish Central Hospital and will include all patients from 2 months up to 18 years of age with seizures admitted to Al-Arish Central Hospital

SUMMARY:
This study will be carried to:

1. Describe the pattern of seizures among cases admitted to Pediatric department at Al-Arish central hospital in North Sinai and compare results with national and international similar studies .
2. Provide the basic descriptive information that is necessary for planning future studies.

DETAILED DESCRIPTION:
A seizure or convulsion is a paroxysmal, time-limited change in motor activity and/or behavior that results from abnormal electrical activity in the brain .

The International League Against Epilepsy (ILAE) and the International Bureau for Epilepsy (IBE) have come to consensus definitions for the terms epileptic seizure and epilepsy, An epileptic seizure is a transient occurrence of signs and/or symptoms due to abnormal excessive or synchronous neuronal activity in the brain but epilepsy is a disorder of the brain characterized by an enduring predisposition to generate epileptic seizures and by the neurobiologic, cognitive, psychological, and social consequences of this condition.

Approximately 4-10% of children experience at least one seizure (febrile or a febrile) in the 1st 16 yr of life, the cumulative lifetime incidence of epilepsy is 3%, and more than half of the cases start in childhood.

Seizure disorder is a general term that is usually used to include any of several disorders, including epilepsy, febrile seizures, and possibly single seizures and symptomatic seizures secondary to metabolic, infectious, or other etiologies (e.g., hypocalcaemia,meningitis).

In the International League Against Epilepsy (ILAE) classification of etiology of epilepsy, idiopathic epilepsy which occur without organic cause, and symptomatic epilepsy that associated with underlying brain disorder that may or may not be genetic .

The definition of epilepsy requires the occurrence of 2 or more unprovoked seizures occur in a time frame of longer than 24 hr .

There are 2 main types of seizures: generalized and focal, focal seizures are those arising within networks of a single cerebral hemisphere and may remain localized or subsequently become more widely distributed.

Generalized seizures rapidly affect both hemispheres as well as both sides of the body even when caused by a "focal" lesion.

Focal (formerly known as partial) seizures are subdivided into simple partial seizures which is refers to focal seizures with no alteration in consciousness and complex partial seizures associated with altered awareness of the surroundings.

Generalized seizures are further subdivided to tonic (sustained contraction), clonic (rhythmic contractions), myoclonic (rapid shock-like contractions, usually<50 msec in duration, that may be isolated or may repeat but usually are not rhythmic), atonic, or astatic (cause avery momentary loss of tone with sudden fall ) Absence seizures (generalized seizures consisting of staring, unresponsiveness, and eye flutter lasting usually for few seconds).

Seizures triggered by fever, defined as febrile seizures, have been for decades a major issue for children in developed countries Epidemiologic studies have led to the division of febrile seizures into 3 groups, as follows:

* Simple febrile seizures
* Complex febrile seizures
* Symptomatic febrile seizures In Simple febrile seizure is single generalized seizure and lasts less than 15 minutes, The child is otherwise neurologically healthy and without neurologic abnormality by examination or by developmental history and not caused by meningitis, encephalitis, or any other illness affecting the brain .

Complex febrile seizure: This seizure is either focal or prolonged (ie, >15 min), or multiple seizures occur in close succession.

Symptomatic febrile seizure: The child has a preexisting neurologic abnormality or acute illness.

Although the outlook for most children with symptomatic seizures or those associated with epilepsy is generally good, seizures may signal a potentially serious underlying systemic or central nervous system (CNS) disorder that requires thorough investigation and management.

Children may have behaviors that are easily mistaken for epileptic Seizures but are not , these include breath-holding spells ,bed wetting ,night terrors ,tics.

Gastroesophageal reflux may cause arching of the back and twisting of the head to the side in infants, which may be mistaken for tonic-clonic seizures, misdiagnosis is frequent (occurring in about 5 to 30% of cases) .

Descriptive epidemiology of pediatric seizures is important for:

First, knowledge of health care utilization is essential for planning and management.

This study will be carried to:

1. Describe the pattern of seizures among cases admitted to Pediatric department at Al-Arish central hospital in North Sinai and compare results with national and international similar studies .
2. Provide the basic descriptive information that is necessary for planning future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 2 months upto 18 years of age with seizures admitted to Al-Arish central Hospital .

Exclusion Criteria:

* No exclusion criteria

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Area of study: Pediatric department at Al-Arish central hospital in North Sinai.
  Descriptive cross sectional hospital based study. Data will be collected from patient using semi structured questionnaire through interview with patient care giver.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-08-24 (Estimated)

PRIMARY OUTCOMES:
Description of the pattern of seizures among cases admitted to Pediatric department at Al-Arish central hospital in North Sinai and compare results with national and international similar studies . | 1 year
  Descriptive cross sectional study Data will be collected from patient using semi structured questionnaire through interview with patient care giver.
  Data will be entered, cleaned and analyzed using statistical software program (SPSS version 20).
  Descriptive statistics will be presented in the form of percentages for qualitative variables and mean and SD for quantitative data.
  Qualitative data will be compared using chi-square test, and quantitative data will be compared using Student's t test, other tests will be used as appropriate .
  P-value will be considered significant if less than0.05 for all statistical tests .

CONTACTS AND LOCATIONS:
Overall Officials: Ehsan mr Saeid, RD, Principal Investigator — Assiut University

REFERENCES:
- [Background] Freeman JM, Tibbles J, Camfield C, Camfield P. Benign epilepsy of childhood: a speculation and its ramifications. Pediatrics. 1987 Jun;79(6):864-8. PMID 3588141
- [Background] Berg AT, Berkovic SF, Brodie MJ, Buchhalter J, Cross JH, van Emde Boas W, Engel J, French J, Glauser TA, Mathern GW, Moshe SL, Nordli D, Plouin P, Scheffer IE. Revised terminology and concepts for organization of seizures and epilepsies: report of the ILAE Commission on Classification and Terminology, 2005-2009. Epilepsia. 2010 Apr;51(4):676-85. doi: 10.1111/j.1528-1167.2010.02522.x. Epub 2010 Feb 26. PMID 20196795
- [Background] Dalbem JS, Siqueira HH, Espinosa MM, Alvarenga RP. Febrile seizures: a population-based study. J Pediatr (Rio J). 2015 Nov-Dec;91(6):529-34. doi: 10.1016/j.jped.2015.01.005. Epub 2015 May 26. PMID 26022778
- [Background] Verity CM, Golding J. Risk of epilepsy after febrile convulsions: a national cohort study. BMJ. 1991 Nov 30;303(6814):1373-6. doi: 10.1136/bmj.303.6814.1373. PMID 1760604
- [Background] Richards CF, Lowe RA. Researching racial and ethnic disparities in emergency medicine. Acad Emerg Med. 2003 Nov;10(11):1169-75. doi: 10.1111/j.1553-2712.2003.tb00599.x. PMID 14597491